CLINICAL TRIAL: NCT06854133
Title: Longitudinal Study Comparing an Italian and a Californian Population of Mentally Ill Offenders: Identification of Forensic Treatment Effectiveness Factors
Brief Title: Factors of Effectiveness in Italian Forensic Treatment
Acronym: REMS FEIFT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Felice Carabellese, MD Full Professor in Forensic Psychiatry, University of Bari
Other Study IDs: REMS FEIFT
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Forensic Psychiatric Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Italian forensic patients: Italian forenisc patients
- Californian Forensic patients: Californian forensic patients

SUMMARY:
Over the last few years, in Italy, the treatment of the mentally ill offender has undergone profound changes following a series of successive legislative interventions. Lastly, Law no. 81 of 30 May 2014 decreed the closure of the 6 active high-security psychiatric hospitals (Ospedali Psichiatrici Giudiziari = OPG), opting for a new model of forensic care.

The new Italian forensic treatment model is essentially community-based, exclusively managed by the health system, with rehabilitation and recovery purposes in the patient's home territory. Due to its characteristics, it is unique in the Western world.

In California, the forensic treatment model is defined by the California Penal Code. The Department of State Hospitals (DSH) oversees the care and security pathways of individuals deemed not criminally responsible by reason of mental disorder (NGRI) or incompetent to stand trial (IST). Care pathways are organized around the secure hospital, with the largest number of beds in high-security hospitals. There are also community-based forensic facilities. The average length of stay is 10 years, two-thirds of which is in the hospital.

The forensic treatment models of the two countries considered are, therefore, very different from each other, each with specific strengths and weaknesses.

Some national data (Catanesi et al, 2019) show that the length of stay in Italian community forensic facilities intended to exclusively accommodate people subject to detention security measures (Residences for the Execution of the Security Measure = REMS) is much shorter than in California.

Furthermore, REMS do not have the same standardization of safety procedures to be followed that is observed in Californian hospitals, whether it concerns structural measures, relational measures, or professional services. There is instead a greater use of psychotherapeutic treatments and rehabilitative and occupational activities. Some experiential data seem to indicate, however, some specific outcome indicators in REMS that suggest greater forensic treatment efficacy compared to Californian forensic hospital facilities.

The differences between the two countries raise important questions about the clinical, therapeutic, and social factors that may be relevant in the forensic recovery process. Understanding the nature of these questions may illustrate a more generalizable understanding of the factors that help people receiving forensic care recover and regain successful social reintegration in a safe manner. Understanding the similarities and contrasts between the two different treatment settings of California and Italy is the primary goal of this study.

Despite the diversity of the forensic models of the two countries considered, we intend to compare the two different treatment realities by enrolling a national sample of Italian forensic patients (Group I) and a sample of forensic patients from the State of California (Group C) of equal numbers, to then follow them both for three years with annual check-ups. Starting from a similar starting time T0 for both patient samples, using the same risk assessment and clinical tools, the same data collection form common to the models of the two countries (containing personal, work, anamnestic, clinical, and judicial data) and a specific treatment evaluation form (quality and type of pharmacological treatment; level of adherence to pharmacological treatment; awareness of the disease and level of adaptation to the treatment measures; quality of the rehabilitation measures chosen; any psychotherapies; family support during the project; commitment to socially useful or work-related activities; economic support), the enrolled patients will be followed for three years starting from time T0 through annual periodic check-ups.

The admission criteria differ between the Californian and Italian systems. However, some patients are similar in diagnosis and type of crime committed. Focusing on patients with similar diagnoses and type of crime committed will allow us to understand the differences that we expect to observe in the different care models. Therefore, for the purposes of comparison, we will focus on patients with diagnoses of psychotic disorder and mental disorder with respect to the crime committed.

DETAILED DESCRIPTION:
The longitudinal study involves the enrolment of all mentally ill offenders, with partial or total mental infirmity, who enter for the first time in Italian forensic care settings (Group I) and Californian hospital forensic facilities (Group C).

For Group I, ex lege reference will be made both to REMS, in the case of custodial security measures, and to other care settings (residential, semi-residential, domicile), in the case of non-custodial security measures. As far as the type of security measure is concerned, both definitive and provisional measures will be considered.

The observation period will be three years from the recruitment period to the target date (time = T0).

All patients will be asked to give written informed consent to participate in the research, in full compliance with the ethical and deontological principles provided; if subject to forms of legal guardianship, the guardian or the Support Administrator will be involved.

Patients in Groups I and C will be monitored for three years from their enrolment with annual check-ups: at twelve months (T1); at twenty-four months (T2); at thirty-six months (T3) or upon discharge from the forensic system, depending on whether this occurs before the expected observation time. At the end of the three years of observation, a structured interview with the Clinical Global Impression - Change (CGI-C) will be conducted with the health workers involved to record their subjective perception of the quality of treatment offered to patients. At the time of discharge, information will be acquired on the patient's subsequent placement and whether discharge is conditional or not. In the event of discharge from the facility involved before the three years of observation expected, the patient, at the time of discharge, will be subjected to the subsequent verification expected with respect to the last one actually carried out, with the same tools provided for by the research protocol. In this case too, the CGI-C will be carried out with the reference health workers, and information will be acquired on the patient's subsequent placement and whether discharge is conditional or not.

The evaluation procedures planned at times T1, T2, and T3 on the enrolled patients must be carried out in a limited period of time (max 2 weeks), the same for all.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* less than MMSE 18 score

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The aim is ultimately to develop reliable and scientifically sound strategies and tools for predicting forensic treatment efficacy and to verify whether and how indications from other countries with different healthcare organizations can also be applied in Italy and vice versa.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Lenght of stay in REMS | from 12.01.2025 to 12.01.2028
  The length of stay in the REMS with unconditional discharge

IPD SHARING:
Plan to Share IPD: Undecided
I have not decided yet